CLINICAL TRIAL: NCT06246006
Title: Functional Characterization of Thrombopoietin/cMPL Receptor Mutations in Myeloproliferative Neoplasia
Acronym: MPL - NPM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2023-1/SC01
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Myeloproliferative Disorder
Keywords: leukemia; neoplasm; polymorphism; thrombocythemia; Thrombopoietin receptor,
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Neoplasms; Thrombocytosis | interventions — Base Sequence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples and bone marrow samples will be taken depending on the clinical management of the patient
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected MPN
  Interventions: Other: Gene sequencing

INTERVENTIONS:
Other: Gene sequencing — Next generation sequencing of candidate genes (JAK2, cMPL, CALR, ASXL1 and NF-E2)

SUMMARY:
The MPL gene is implicated in two groups of hematological pathologies: congenital amegakaryocytic thrombocytopenia (CAMT) and Phi negative myeloproliferative neoplasia (MPN). Fifty germline mutations have been identified in CAMT, yet only a dozen activating mutations have been described in MPN. Most are somatic, distributed mainly in the transmembrane (TM) and juxtamembrane (JM) domains. However, a few rare germline mutations located in the extracellular domain (ECD) have also been reported: K39N, R102P and P106L.

Next generation sequencing technology has been used to study the complete MPL gene, identifying numerous variants, most of unknown significance. The study investigators have a series comprising 41 variants of unknown significance, whose allelic frequencies suggest a germline origin for 80% of them. Their distribution within the MPL gene is similar to that of inactivating mutations, except that they were discovered in the context of suspected myeloproliferative disease. Characterizing the activity of these variants would confirm the diagnosis of MPN, opening the door to specific treatment (cytoreductive, JAK2 inhibitor or interferon). It also has an important prognostic value, particularly in the case of MPN, for which life expectancy varies from 5 to 7 years, with terminal progression to acute myeloid leukemia (AML in 15 to 20% of cases) or bone marrow failure.

Using a battery of functional assays, this study aims to characterize these variants.

ELIGIBILITY:
Inclusion Criteria:

• Patient with suspected MPN

Exclusion Criteria:

• Patient with variant of cMPL already described in the literature.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with suspected MPN screened at CHU Nîmes
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Growth of cultured cells with site-directed mutagenesis of identified variants in the presence of thrombopoietin | Day 0
  Thrombopoietin concentration curve
Ability of cultured cells with site-directed mutagenesis of identified variants to activate the MPL - JAK2 pathway | Day 0
  STAT5 Luciferase reporter system
Ability of cultured cells with site-directed mutagenesis of identified variants to phosphorylate proteins in the MPL - JAK2 pathway | Day 0
  Western blot of JAK2, STAT (3 and 5) AKT, ERK1 /2 proteins

CONTACTS AND LOCATIONS:
Overall Officials: Serge Carillo, Principal Investigator — CHU de Nimes
Locations (1):
- CHU de Nîmes, Nîmes, France